CLINICAL TRIAL: NCT03068273
Title: Managing Type 1 and High Risk Type 2 Diabetes in the Hospital Setting: Glucose as a Vital Sign
Acronym: CGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Whittier Diabetes Institute (Other)
Responsible Party: Principal Investigator, Athena Philis-Tsimikas, Corporate Vice President, Scripps Whittier Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-6878
Record Dates: First submitted 2016-10-12; First posted 2017-03-01 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Hospitalization
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention (Experimental): For type 2 patients in the intervention group, CGM data will be viewed real-time.
  Interventions: Device: Real-time CGM data
- Control (Experimental): For type 2 patients in the control group, CGM data is blinded to all and only gathered for comparison purposes to intervention group.
  Interventions: Device: Real-time CGM data

INTERVENTIONS:
Device: Real-time CGM data

SUMMARY:
This program will provide patients with type 1 and high risk type 2 diabetes the safest hospitalization by using wireless continuous glucose monitoring devices (CGM) to track their glucose parameters in real-time similar to other continuously monitored vital signs. The CGM will inform a team of health professionals who will monitor the patients' progress, communicate recommendations, and be available for discussion when recommended targets are not achieved. Health teams will utilize sensor results in addition to existing electronic medical records data to evaluate progress and manage care.

DETAILED DESCRIPTION:
All patients with type 1 or type 2 diabetes who meet study criteria will be invited to participate in the study. All patients included in the study will be followed by an advanced practice diabetes nurse for glucose management during their hospitalization. All patients included in the study will receive a CGM. Patients with type 2 diabetes will be randomized to control (blinded CGM glucose values to APN, care team and researchers) or intervention (CGM blood glucose values will be used to aid with glucose management during the hospitalization). In addition, a research only supplemental order set will be implemented for all study participants. The order set focuses on any glucose point of care test that is between 70-79 mg/dL or ≥ 250 at bedtime or before the 4 am usual care blood glucose check. The goal is to prevent hypoglycemia and hyperglycemia for all study patients. The advanced practice diabetes nurse will work with the physician in charge of the patient's care as well as the patient's care team.

ELIGIBILITY:
Inclusion Criteria:

* Expected length of hospital stay of at least 48 hours
* One of the following:

  1. Diagnosed with diabetes type 1 OR
  2. Diagnosed with diabetes type 2, with an HbA1c > 8% or 3 point-of-care blood glucose (POC) > 200, and requiring insulin during this hospitalization.
* Literate in English or Spanish

Exclusion Criteria (not all listed):

* Pregnant or post-partum
* Patient admitted to OB unit
* Patient in ICU or with insulin drip
* Known allergy to adhesives
* Anticipated CT/MRI/diathermy procedure within 48 hours from admission (patients with a planned operation within 48 hours from admission may be included in the study post operation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Athena Philis-Tsimikas, MD, Principal Investigator — Scripps Whittier Diabetes Institute
Locations (1):
- Scripps Whittier Diabetes Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortmann AL, Spierling Bagsic SR, Talavera L, Garcia IM, Sandoval H, Hottinger A, Philis-Tsimikas A. Glucose as the Fifth Vital Sign: A Randomized Controlled Trial of Continuous Glucose Monitoring in a Non-ICU Hospital Setting. Diabetes Care. 2020 Nov;43(11):2873-2877. doi: 10.2337/dc20-1016. Epub 2020 Aug 27. PMID 32855160

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients in the intervention group, CGM data will be viewed real-time.
  Real-time CGM data
- Control: Patients in the control group, CGM data is blinded to all and only gathered for comparison purposes to intervention group.
  Real-time CGM data
- Observational T1D: Hospitalized patients with T1D placed on a CGM
Period: Overall Study
Arm/Group | Intervention | Control | Observational T1D
Started | 57 | 53 | 47
Completed | 57 | 53 | 47
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: For type 2 patients in the intervention group, CGM data will be viewed real-time.
  Real-time CGM data
- Control: For type 2 patients in the control group, CGM data is blinded to all and only gathered for comparison purposes to intervention group.
  Real-time CGM data
- Observational T1D: For type 1 patients in the observational group, CGM data will be viewed real-time.
  Real-time CGM data
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Observational T1D | Total
Number analyzed (Participants) | 57 | 53 | 47 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.88 (14.01) | 60.94 (12.37) | 43.6 (12.73) | 61.94 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 22 | 82
  Male | 27 | 23 | 25 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Missing data at hospital admission.
  Participants
    number analyzed (Participants) | 57 | 52 | 47 | 156
    Hispanic or Latino | 39 | 42 | 16 | 97
    Not Hispanic or Latino | 18 | 10 | 31 | 59
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 57 | 53 | 47 | 110
Type 2 Diabetes Duration [Mean (Standard Deviation); unit: years] — Population: Missing data at hospital admission. Explanation: Data not assessed in T1D observational arm
  years
    number analyzed (Participants) | 56 | 51 | 0 | 107
    (all) | 16.23 (9.74) | 18.51 (12.04) |  | 17.37 (10.89)
HbA1c at Hospital Admission [Median (Inter-Quartile Range); unit: percentage] — Population: HbA1c was missing on patients
  percentage
    number analyzed (Participants) | 49 | 44 | 47 | 140
    (all) | 9.5 [7.6 to 11.1] | 8.65 [7.68 to 10.53] | 9.5 [8.1 to 11.2] | 9.075 [7.6 to 11.1]
Point of Care (POC) Blood Glucose Testing at Hospital Admission [Median (Inter-Quartile Range); unit: mg/dL] — Population: Missing data at hospital admission.
  mg/dL
    number analyzed (Participants) | 55 | 52 | 47 | 154
    (all) | 261 [213 to 315] | 245.5 [196.5 to 298.25] | 334.00 [183.0 to 568.0] | 253.25 [196.5 to 315]
Serum Creatinine at Hospital Admission [Median (Inter-Quartile Range); unit: mg/dL] — Population: Range not determined in this T1D observational arm
  mg/dL
    number analyzed (Participants) | 57 | 53 | 0 | 110
    (all) | 1.00 [0.60 to 2.10] | 1.00 [0.70 to 1.90] |  | 1.00 [0.60 to 2.10]
BMI [Median (Inter-Quartile Range); unit: kg/m2] — Population: Missing data at hospital admission. Explanation: BMI not collected in this T1D observational arm
  kg/m2
    number analyzed (Participants) | 56 | 48 | 0 | 104
    (all) | 29.9 [25.02 to 33.40] | 30.65 [25.27 to 36.20] |  | 30.27 [25.02 to 36.20]

OUTCOME MEASURES:

1. Primary Outcome: Type 2 Diabetes Blood Glucose Time in Range (70-180 mg/dL)
Description: Percentage of time a person's blood glucose level stays within a specific range of 70-180 mg/dL
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: percentage of time during CGM use
Groups:
- Observational T1D: For type 1 patients in the observational group, real-time CGM data was collected.
Arm/Group | Intervention | Control | Observational T1D
Number analyzed (Participants) | 57 | 53 | 47
percentage of time during CGM use | 25.31 [11.78 to 42.97] | 19.89 [3.34 to 40.09] | 26.04 [10.40 to 49.57]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.1460, Regression, Linear
Statistical Analysis 2: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear
Statistical Analysis 3: Comparison: Intervention vs Control; Test type: Superiority; p < 0.05, Regression, Linear; Mean Difference (Net) = 6.338, Standard Error of Mean 4.331

2. Primary Outcome: Type 2 Diabetes Blood Glucose Time in Range (70-200 mg/dL)
Description: Percentage of time a person's blood glucose level stays within a specific range on 70-200 mg/dL
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: percentage of time during CGM use
Arm/Group | Intervention | Control | Observational T1D
Number analyzed (Participants) | 57 | 53 | 47
percentage of time during CGM use | 42.82 [25.66 to 58.53] | 33.38 [10.90 to 55.74] | 33.57 [18.19 to 61.54]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.0615, Regression, Linear; Mean Difference (Net) = 9.141, Standard Error of Mean 4.838

3. Primary Outcome: Type 2 Diabetes Blood Glucose Time in Range (70-250 mg/dL)
Description: Percentage of time a person's blood glucose level stays within a specific range on 70-250 mg/dL
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: percentage of time during CGM use
Arm/Group | Intervention | Control | Observational T1D
Number analyzed (Participants) | 57 | 53 | 47
percentage of time during CGM use | 72.83 [59.03 to 83.57] | 63.95 [31.25 to 77.95] | 65.97 [44.10 to 87.00]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.0404, Regression, Linear; Mean Difference (Net) = 11.257, Standard Error of Mean 4.775

4. Secondary Outcome: Percentage Time in Hypoglycemia (<70 mg/dL)
Description: Percentage of time a person's blood glucose level stays within a specific range < 70 mg/dL
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: percentage of time during CGM use
Arm/Group | Intervention | Control | Observational T1D
Number analyzed (Participants) | 57 | 53 | 47
percentage of time during CGM use | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.2680, Regression, Linear; Mean Difference (Net) = 0.155, Standard Error of Mean 0.354

5. Secondary Outcome: Percentage Time in Hyperglycemia (>250 mg/dL)
Description: Percentage of time a person's blood glucose level stays within a specific range > 250 mg/dL
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: percentage of time during CGM use
Arm/Group | Intervention | Control | Observational T1D
Number analyzed (Participants) | 57 | 53 | 47
percentage of time during CGM use | 27.00 [16.01 to 40.97] | 32.96 [20.40 to 68.75] | 34.04 [5.90 to 55.90]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.0403, Regression, Linear; Mean Difference (Net) = -11.412, Standard Error of Mean 4.839

ADVERSE EVENTS:
Time Frame: Length of time on study over a 2-year period
Groups:
- Intervention: Patients with T2D in the intervention group, CGM data will be viewed real-time.
  Real-time CGM data
- Control: Patients with T2D in the control group, CGM data is blinded to all and only gathered for comparison purposes to intervention group.
  Real-time CGM data
Arm/Group | Intervention | Control | Observational T1D
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/53 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/53 | 0/47
Other Adverse Events (participants affected / at risk) | 0/57 | 0/53 | 0/47

LIMITATIONS AND CAVEATS:
The control group was not considered ethical for the T1D arm; therefore, no comparison data was available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT03068273/Prot_SAP_000.pdf